CLINICAL TRIAL: NCT05104294
Title: Correlation Between Optical Coherence Tomography Angiography and Photopic Negative Response in Patients With Primary Open Angle Glaucoma
Brief Title: Correlation Between Optical Coherence Tomography Angiography and Photopic Negative Response in Patients With Glaucoma
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelshafy, Lecturer of Ophthalmology, Benha University
Other Study IDs: RC-9-11-01
Record Dates: First submitted 2021-10-20; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Open Angle Glaucoma
Keywords: Open angle glaucoma; Optical coherence Tomography; Photopic negative response
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- mild Primary Open Angle Glaucoma group (Group I): 28 eyes of 16 patients with mild primary open angle glaucoma as group I.
  Interventions: Diagnostic Test: Optical Coherence Tomography- Angiography; Diagnostic Test: Photopic negative response
- moderate to severe Primary Open Angle Glaucoma group (Group II): 44 eyes of 24 patients with moderate to severe primary open angle glaucoma as group II.
  Interventions: Diagnostic Test: Optical Coherence Tomography- Angiography; Diagnostic Test: Photopic negative response
- Control Group: 80 eyes of 40 healthy subjects as control group.
  Interventions: Diagnostic Test: Optical Coherence Tomography- Angiography; Diagnostic Test: Photopic negative response

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography- Angiography — Peripapillary retinal nerve fiber layer thickness, ganglion cell complex, superficial and deep capillary plexus vessel density were measured.
  Other Names: OCT-A
Diagnostic Test: Photopic negative response — Both the implicit time and amplitude of PhNR were recorded.
  Other Names: PhNR

SUMMARY:
Open angle glaucoma (OAG) is considered a common cause of irreversible vision loss worldwide. It is an optic neuropathy associated with progressive loss and degeneration of the retinal ganglion cell layer (RGC) and its axons (retinal nerve fiber layer; RNFL), which lead to neuroretinal rim excavation and corresponding visual field defects.

DETAILED DESCRIPTION:
Open angle glaucoma (OAG) is considered a common cause of irreversible vision loss worldwide. It is an optic neuropathy associated with progressive loss and degeneration of the retinal ganglion cell layer (RGC) and its axons (retinal nerve fiber layer; RNFL), which lead to neuroretinal rim excavation and corresponding visual field defects.

OCT Angiography (OCTA) is a promising tool for diagnosing and monitoring glaucomatous patients. It can evaluate glaucomatous damage and assess the ganglion cells' health by measuring blood flow within the optic nerve and the retina Correlation between vascular , structural and functional changes of the peripapillary retinal nerve fiber (RNFL) and macular/ganglion cell complex (GCC) can lead to early detection of glaucomatous changes.

ELIGIBILITY:
Inclusion Criteria:

* Age of 30 years or older for both control and glaucoma groups.
* Spherical equivalent (SE) between -2 and +2 D.
* No history of previous eye surgery, trauma, or systemic diseases.

Exclusion Criteria:

* Spherical equivalent greater than +/- 2.00 diopters (D).
* Media opacity as (cataract or corneal scar).
* Any history of ocular surgeries or trauma.
* Optic nerve anomaly or other retinal diseases.
* Unreliable visual field tests (33% fixation losses, false positive, and false- negative results).

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: One hundreds fifty-two eyes of 76 participants were included in this study, with the participants recruited from the outpatient glaucoma clinic of Benha University Hospital, EGYPT.
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2020-02-02 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Correlation between vascular, structural and functional changes of the peripapillary retinal nerve fiber and macular ganglion cell complex in patients with open angle glaucoma. | Immediately after OCTA and electroretinogram diagnostic tests for each eye.
  Correlation between RNFL thickness and GCC measured by OCT-A with implicit time and amplitude of Photopic Negative Response (PhNR) measured by electroretinogram.

SECONDARY OUTCOMES:
Assess the validity of OCTA parameters and PhNR in early detection of glaucoma changes. | Immediately after OCTA and electroretinogram diagnostic tests for each eye.
  Changes in the parameters were measured by OCT-A as Superficial and deep vessel Density.

CONTACTS AND LOCATIONS:
Overall Officials: Marwa A Tabl, MD, Study Chair — Benha University
Locations (1):
- Benha University, Banhā, Benha, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tabl AA, Tabl MA. Correlation between OCT-angiography and photopic negative response in patients with primary open angle glaucoma. Int Ophthalmol. 2023 Jun;43(6):1889-1901. doi: 10.1007/s10792-022-02588-9. Epub 2022 Nov 28. PMID 36441346